CLINICAL TRIAL: NCT03657927
Title: A Comparison of McGrath® MAC Versus C-MAC® Videolaryngoscopes in Morbidly Obese Patients Undergoing Bariatric Surgery: A Randomized, Controlled Clinical Trial
Brief Title: A Comparison of McGrath MAC Versus C-MAC Videolaryngoscopes in Morbidly Obese Patients
Acronym: mcgrath&cmac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sedat AKBAS, Asst. Prof. Dr. Sedat Akbas, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: sedatakbas3
Record Dates: First submitted 2018-08-07; First posted 2018-09-05 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Difficult Intubation; Morbid Obesity; Videolaryngoscopy
Keywords: Morbidly Obese; Difficult Airway Management; Videolaryngoscopy
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- C-MAC Videolaryngoscope (Active Comparator): Morbidly obese patients intubated with C-MAC Videolaryngoscope
  Interventions: Device: C-MAC videolaryngoscope; Device: McGrath MAC videolaryngoscope
- McGrath MAC Videolaryngoscope (Active Comparator): Morbidly obese patients intubated with McGrath MAC Videolaryngoscope
  Interventions: Device: C-MAC videolaryngoscope; Device: McGrath MAC videolaryngoscope

INTERVENTIONS:
Device: C-MAC videolaryngoscope — An intubating device that is used for endotracheal intubation. Endotracheal intubation was applied by anesthesiologist with C-MAC videolaryngoscope.
Device: McGrath MAC videolaryngoscope — An intubating device that is used for endotracheal intubation. Endotracheal intubation was applied by anesthesiologist with McGrath MAC videolaryngoscope.

SUMMARY:
Along with the technological advances in medicine, videolaryngoscope is the most commonly preferred technique for intubation of expected difficult airway management such as morbidly obese patients. In this prospective controlled clinical study, the purpose is to compare C-MAC videolaryngoscope and McGrath MAC videolaryngoscope in respect to duration of intubation, haemodynamic response, and complications related intubation of morbidly obese patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
It is very important for anesthesiologists to evaluate and make the airway safe in order to start and continue surgical operations. Endotracheal intubation has many important reasons such as ensuring airway control safely during surgical procedure, increasing the depth of anesthesia, need interventions for surgical or anesthetic complications, reduction of dead space, reduction of respiratory effort and prevention of aspiration risk.

Mask ventilation and tracheal intubation in morbidly obese patients can be difficult with the anatomical changes caused by obesity. Reduced functional residual capacity in morbidly obese patients makes it difficult to maintain peripheral oxygen saturation at normal limits. Videolaryngoscope, developed in recent years and beginning to take place in the algorithms, facilitate difficult airway management and hence intubation.

The use of videolaryngoscope in patients with difficult intubation such as morbid obesity, has been frequently reported in the literature. McGrath videolaryngoscope has a high-resolution video camera, a length-adjustable angle blade, and a light source at the tip of the blade. At the same time, the C-MAC videolaryngoscope is another advanced videolaryngoscope with a better quality video and camera system and improves the performance of videolaryngoscope with some technological changes.

In this prospective controlled clinical study, the purpose is to compare C-MAC videolaryngoscope and McGrath MAC videolaryngoscope in respect to duration of intubation, haemodynamic response, and adverse events associated with intubation of morbidly obese patients undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology score III,
* 18-65 years,
* BMI> 40

Exclusion Criteria:

* American Society of Anesthesiology IV,
* Under 18 years,
* Over 65 years,
* Under BMI<40
* Obstetric patients,
* Uncontrolled cerebrovascular disease,
* Patients who refused written informed consent forms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-08 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Time to intubation | From beginning of holding videolaryngoscope to seeing two meaningful end-tidal carbon dioxide levels up to 3 minutes
  Time to intubation was defined as the time from when the anesthesiologist picked up the videolaryngoscope to when the anesthesiologist successfully placed the endotracheal tube through the vocal cords

SECONDARY OUTCOMES:
Heart Rate | From beginning of Anesthesia induction to 5th minutes of intubation
  Heart Rate
Mean Arterial Pressure | From beginning of Anesthesia induction to 5th minutes of intubation
  Mean Arterial Pressure
Adverse Events | During the first 24 hour postoperatively
  Bleeding in the mouth, edema in the mouth, burst of intubation tube cuff, external laryngeal press, presence of head position change, laryngospasm, hypoxia, hoarseness, throat ache

CONTACTS AND LOCATIONS:
Overall Officials: Sedat Akbas, Study Director — Inonu University Medical Faculty
Locations (1):
- Sedat AKBAS, Malatya, Türkiye-Türkçe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaszynski T. Clinical experience with the C-Mac videolaryngoscope in morbidly obese patients. Anaesthesiol Intensive Ther. 2014 Jan-Mar;46(1):14-6. doi: 10.5603/AIT.2014.0003. PMID 24643921
- [Background] Taylor AM, Peck M, Launcelott S, Hung OR, Law JA, MacQuarrie K, McKeen D, George RB, Ngan J. The McGrath(R) Series 5 videolaryngoscope vs the Macintosh laryngoscope: a randomised, controlled trial in patients with a simulated difficult airway. Anaesthesia. 2013 Feb;68(2):142-7. doi: 10.1111/anae.12075. Epub 2012 Nov 5. PMID 23121470

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT03657927/Prot_SAP_001.pdf